CLINICAL TRIAL: NCT00842998
Title: A Phase II, Randomized Trial With Single Agent Trastuzumab or Lapatinib in Patients With Metastatic HER2-Overexpressing Breast Cancer
Brief Title: Efficacy Study of Single Agent Trastuzumab or Lapatinib to Treat HER2-Overexpressing Breast Cancer
Acronym: HERLAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Ordine Mauriziano di Torino (Other)
Responsible Party: Prof. Massimo Aglietta / Dr Filippo Montemurro, I.R.C.C. - A.O. Ordine Mauriziano di Torino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080331 - HERLAP; EudraCT No: 2008-001916-18
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; HER2; Trastuzumab; Lapatinib; HER2 gene-amplification
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - Trastuzumab (Experimental): Day1 Week1: 8 mg/kg iv in 90 min. Following 1st week: 2 mg/kg once/weekly for 8 weeks
  Interventions: Drug: Trastuzumab or Lapatinib
- 2 - Lapatinib (Experimental): 1500 mg/die orally
  Interventions: Drug: Trastuzumab or Lapatinib

INTERVENTIONS:
Drug: Trastuzumab or Lapatinib — Trastuzumab: loading dose 8 mg/kg iv in 90 min.followed by weekly doses of 2 mg/kg Lapatinib: 1500 mg/die orally

SUMMARY:
This study will evaluate the activity of single agent trastuzumab or lapatinib in patients not previously treated for HER-2 positive (FISH positive) metastatic breast cancer. A companion biological study will assess factors correlated with sensitivity or resistance to either one of the compounds

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-75 years
* Histologically or cytologically confirmed metastatic disease.
* HER2-Overexpression proven by Fluorescence in Situ Hybridization (FISH).
* Availability of paraffin-embedded block of either primitive tumor and/or biopsy of metastases.
* No prior chemotherapy for metastatic or locally advanced disease. Patients with hormone receptor (oestrogen and/or progesterone) positive breast cancer can be eligible provided that they had received only ONE line of hormonal therapy for metastatic disease.
* For patients undergoing hormonal therapy for metastatic disease, disease progression must be confirmed according to RECIST criteria.
* At least 20% increase in the sum of longest diameters, OR
* Evidence of new metastatic lesions or progression of pre-existing non-target lesions.
* Presence of at least one monodimensionally measurable lesion. Patients without clinically or radiologically proven evidence of disease are not eligible.
* Patients with exclusively skin disease are eligible, provided that the disease evolution under treatment can be photographically documented.
* Patients with involvement of NCS, besides presence of measurable lesions, are eligible provided that:

  * Brain lesion/s has/have been radically resected;
  * Brain lesion/s has/have obtained complete remission following radiation therapy. Complete remission must be documented by TC or RMN.
* At least 4-week interval from end of radiotherapy, hormono- or immunotherapy and enrollment in this study.
* ECOG PS </= 2 and life expectancy of at least 6 months.
* Liver metastases involving < 30% of liver volume.
* Adequate hematopoietic, liver and renal function
* Written informed consent.
* Patients with childbearing potential must have negative pregnancy test and must use adequate contraceptive measures during treatment.
* Prior treatment with Trastuzumab as adjuvant therapy is permitted provided that it was completed at least 12 months prior enrollment in this study.

Exclusion Criteria:

* Prior chemotherapy for metastatic disease.
* Active pregnancy or breastfeeding.
* Previous treatment with Lapatinib.
* Previous therapy with mono- or policlonal antibodies for metastatic disease.
* Patients with bone involvement or pleural effusion/ascites as unique localization of disease.
* Patients with dyspnea due to presence of disease (lymphangitis) or requiring oxygen therapy.
* Patients with clinically evident hearth disease and/or active infectious diseases.
* Patients with not resected or not irradiated brain and/or leptomeningeal metastases.
* Prior or actual concurrent neoplasms, with the exception of adequately treated carcinoma della cervice uterina and basal cell or squamocellular carcinoma of the skin.
* Patients with uncontrolled serious illnesses that may compromise the compliance of the patient to the treatment.
* Previous allergic reactions towards any excipient in the composition of Trastuzumab or Lapatinib.
* Use of any experimental drug within 4 weeks prior initiation of study treatment.
* Women with childbearing potential who refuse to use adequate contraceptive measures.
* Patients unable to give written informed consent or are not compliant with treatment.
* Patients with great tumor involvement (> 30% dof hepatic volume, etc).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically definite response confirmed by CT or MRI | 8 weeks

SECONDARY OUTCOMES:
Time to Progression (TTP) and duration of response in patients treated with Trastuzumab | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Aglietta, Full Professor, MD, Study Chair — University of Turin Medical School at AO Ordine Mauriziano di Torino; Filippo Montemurro, MD, Principal Investigator — AO Ordine Mauriziano di Torino
Locations (4):
- Italy (4):
  - U.O. Oncologia Medica - Ospedale San Luigi, Orbassano, Torino
  - Institute for Cancer Research and Treatment (I.R.C.C.), Candiolo , Torino
  - U.O. Oncologia Medica, Cuneo
  - U.O. Oncologia Medica - COES Molinette, Torino